CLINICAL TRIAL: NCT02567838
Title: LIdocaine Gel Versus Plain Lubricating Gel for Pain Reduction During Transrectal Sonography (LIPS)
Brief Title: Lidocaine Gel During Transrectal Sonography
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2015-08-022
Record Dates: First submitted 2015-10-01; First posted 2015-10-05 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Gynecologic Diseases
MeSH Terms: conditions — Genital Diseases, Female | interventions — chlorhexidine gluconate, lidocaine drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine gel (Experimental): Instillagel (2% lidocaine) was administered rectally prior to probe insertion.
  Interventions: Drug: Lidocaine gel
- Placebo (Placebo Comparator): Placebo (Aquagel) was administered rectally prior to probe insertion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine gel — Instillagel (2% lidocaine) was administered rectally prior to probe insertion.
  Other Names: Instillagel
  Arms: Lidocaine gel
Drug: Placebo — Placebo (Aquagel) was administered rectally prior to probe insertion.
  Other Names: Aquagel
  Arms: Placebo

SUMMARY:
The aim of this clinical trial is to evaluate the use of topical lidocaine gel in reducing pain associated with transrectal ultrasonography (TRS) in gynecologic field.

DETAILED DESCRIPTION:
TRS is the common procedure to diagnose or exclude gynecologic disease in virgin women. This procedure can be associated with significant pain, both on insertion of the ultrasound probe as well as on manipulating the probe. The investigators evaluated a new technique for pain relief during TRS. In all, 80 consecutive subjects undergoing TRS at obstetric and gynecologic department were randomized to receive either lidocaine gel(Instillagel) or placebo(Aquagel) rectally prior to probe insertion. The pain encountered before, during, and after the procedure was graded by the patient on a 10-point visual analogue score. The gel-associated side effect was also evaluated by phone survey after 2 day of procedure. The aim of this clinical trial is to evaluate the use of topical lidocaine gel in reducing pain associated with transrectal gynecologic ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* All virgin women who were scheduled to undergo transrectal sonography invited to participate.

Exclusion Criteria:

* Allergy to lidocaine or other local anesthetics;
* Patients with a chronic pain condition for which they were taking daily pain medications of any kind.
* A bleeding diathesis and/or anticoagulant treatment;
* Underlying anal or rectal diseases such as symptomatic hemorrhoid, anal fissure, fistulae or anal stricture;
* An inability to rate a visual analogue scale

Ages: 15 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Pain assessed by a 10-point visual analogue score | the day of the procedure (transrectal sonography)

SECONDARY OUTCOMES:
Number of participants with gel-associated side effect | 2 days after the procedure (transrectal sonography)
  Information on side effect was collected by phone survey

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, MD PhD, Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No